CLINICAL TRIAL: NCT04406701
Title: Impact of the Health Crisis and the Economic Situation in Lebanon on the Eating Habits of Lebanese Nurses.
Brief Title: Ceres: Eating Habits Among Lebanese Nurses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Paris 13 (Other)
Responsible Party: Principal Investigator, Rita Nohra, Principal Investigator, University of Paris 13
Other Study IDs: Ceres:observational study
Record Dates: First submitted 2020-05-19; First posted 2020-05-28 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Eating Habits; Nurses
MeSH Terms: conditions — Feeding Behavior | interventions — At4g23840 protein, Arabidopsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ceres — This will be a self-administered survey on eating habits and their relationship to coping strategies and economic level among nurses.

SUMMARY:
The main objective of this research is to study the impact of the health crisis and the economic situation in Lebanon on the eating habits of Lebanese nurses.

It is a descriptive, study among Lebanese nurses working in hospitals. It will be a self-administered survey on eating habits and their relationship with coping strategies and economic level among nurses. Analyses will be carried out using Statistical Package for Social Sciences (SPSS) 21 software.

The results of this study will make a unique and collective contribution to the areas of nursing management and the prevention of eating disorders among nurses.

ELIGIBILITY:
Inclusion Criteria:

* nurses working in hospitals

Exclusion Criteria:

* Maternity leave
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: nurses working in hospitals
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Crowding index | 2 month
  Measure of socio-economic status widely used in socio-economic surveys, it will be calculated as the number of people living in the same house/number of rooms in the house (excluding kitchen and bathrooms). An index > 1 indicates an overcrowded house with few economic resources.
Food Frequency Questionnaire (FFQ) | 2 month
  questionnaire used to obtain frequency and, in some cases, portion size information about food and beverage consumption over a specified period of time, typically the past month or year
Brief Cope | 2 month
  The Brief-COPE is a self-assessment questionnaire designed to measure effective and ineffective ways of coping with a stressful life event.